CLINICAL TRIAL: NCT02223390
Title: Improving the Health of South African Women With Traumatic Stress in HIV Care
Brief Title: Improving the Health of South African Women With Traumatic Stress in HIV Care (C0147)
Acronym: ImpACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Cape Town (Other)
Responsible Party: Principal Investigator, Kathleen Sikkema, Professor, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0979; R34MH102001 (NIH)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: HIV; Trauma Exposure
Keywords: South Africa; HIV; Mental health; Trauma; Women
MeSH Terms: conditions — Psychological Well-Being; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mental health treatment (Experimental): The experimental condition, ImpACT, was developed in the pilot phase of the study. The intervention will be 4 sessions of individual psychological treatment related to stress, coping, and HIV adherence, followed by three group sessions. Sessions will follow an intervention manual and be delivered by a psychiatric nurse (or equivalent nonspecialist in mental health) who is supervised by a trained clinical psychologist.
  Interventions: Behavioral: Improving AIDS Care after Trauma (ImpACT)
- Standard of Care (No Intervention): Participants in standard of care will receive the three-session adherence counseling delivered in the clinic, along with referrals for trauma treatment.

INTERVENTIONS:
Behavioral: Improving AIDS Care after Trauma (ImpACT)
  Arms: Mental health treatment

SUMMARY:
In this study, the investigators propose to develop Improving AIDS Care after Trauma (ImpACT), an intervention based on theories of stress and coping and evidence-based treatment for traumatic stress. The intervention will target women in South Africa who have histories of sexual trauma and are newly initiating antiretroviral therapy (ART) in order to reduce avoidant coping and traumatic stress, improve care engagement, and reduce HIV risk behaviors.

DETAILED DESCRIPTION:
HIV-infected women in South Africa report high rates of sexual trauma, which negatively impacts their mental health and potentially influences engagement in HIV care (retention in care and adherence to antiretroviral therapy) and risk behaviors. Addressing the traumatic stress resulting from sexual trauma could improve these HIV-related outcomes, which in turn may prevent HIV transmission through suppression of the virus and reduction in HIV risk behaviors. Intervention research among HIV-infected populations with trauma histories in the U.S. demonstrates that a coping approach, particularly one that reduces the use of avoidant coping strategies, is efficacious in reducing traumatic stress and improving health behaviors. Although South Africa faces dual epidemics of HIV and sexual violence, trauma treatment has not been well-integrated into the HIV care setting. The proposed 3-year study will develop and pilot test an intervention called ImpACT (Improving AIDS Care after Trauma) to reduce avoidant coping, traumatic stress, and risk behaviors, and increase engagement in care. The intervention will take place in a public ART clinic and will target women during the critical period when they initiate ART in order to maximize the impact on engagement in care. Qualitative data collection with staff, providers, and HIV-infected female patients at the study clinic will elicit feedback on the content and delivery of ImpACT and key aspects of the study protocol. ImpACT will then be piloted with 60 women who are new ART enrollees with a history of sexual trauma and elevated traumatic stress. Participants will be randomized to the control condition (standard of care, or SoC: 3 adherence counseling sessions required of all patients initiating ART at the clinic) or the intervention condition (SoC + ImpACT), and will complete assessments at baseline, 3, and 6 months post-randomization, with care engagement data extracted from medical records at the end of the study period. The study has three specific aims: 1) to develop a brief and scalable coping intervention for delivery in the South African HIV care setting for women with sexual trauma histories; 2) to establish the methodological details of an experimental protocol for a robust randomized control trial; and 3) to pilot test the ImpACT intervention with 60 HIV-infected women with histories of sexual trauma who are initiating ART in order to determine feasibility and acceptability in the HIV care setting, and explore the impact on avoidant coping, traumatic stress, engagement in care, and HIV risk behaviors. The goal at the completion of this study is to have a structured intervention curriculum that is culturally relevant for HIV infected women in South Africa, a full experimental protocol that is appropriate for the South African care setting, and data on feasibility, acceptability, and target outcomes. These products can be leveraged to inform an R01 application for rigorous evaluation of the ImpACT intervention. We are confident that this developmental work will significantly enhance the probability of success of a larger randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected women who are newly initiating ART at the study clinic
* History of sexual trauma
* Meets criteria for traumatic stress

Exclusion Criteria:

* Immediate suicide risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Sikkema, PhD, Principal Investigator — Duke University (Currently at Columbia University)
Locations (1):
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sikkema KJ, Mulawa MI, Robertson C, Watt MH, Ciya N, Stein DJ, Cherenack EM, Choi KW, Kombora M, Joska JA. Improving AIDS Care After Trauma (ImpACT): Pilot Outcomes of a Coping intervention Among HIV-Infected Women with Sexual Trauma in South Africa. AIDS Behav. 2018 Mar;22(3):1039-1052. doi: 10.1007/s10461-017-2013-1. PMID 29270789

RESULTS

PARTICIPANT FLOW:
Groups:
- Mental Health Treatment: The experimental condition, ImpACT, was developed in the pilot phase of the study. The intervention will be 4 sessions of individual psychological treatment related to stress, coping, and HIV adherence, followed by three group sessions. Sessions will follow an intervention manual and be delivered by a psychiatric nurse (or equivalent nonspecialist in mental health) who is supervised by a trained clinical psychologist.
  Improving AIDS Care after Trauma (ImpACT)
Period: Overall Study
Arm/Group | Mental Health Treatment | Standard of Care
Started | 32 | 32
Completed | 23 | 28
Not Completed | 9 | 4
Not completed — Lost to Follow-up | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mental Health Treatment | Standard of Care | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (6.6) | 29.0 (8.4) | 29.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 32 | 64
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 32 | 32 | 64
PTSD Symptoms (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — Self-report, measured by the PTSD checklist, civilian version (PCL-5). 20-item self-report questionnaire. Participants were asked to indicate the extent to which they were bothered by problems experienced in the past month in relation to a traumatic experience of abuse or act of violence (0 = not at all to 4 = extremely). Total severity score (range: 0-80; higher scores indicating higher symptom severity, >= 33 indicating PTSD) and subscale totals (Avoidance - Cluster C, range: 0-8; and Hyperarousal - Cluster E, range: 0-24) were examined.
  units on a scale
    PCL - total symptom severity score | 43.28 (21.94) | 30.72 (20.27) | 37.00 (21.89)
    PCL - Cluster C Avoidance | 4.53 (2.93) | 3.03 (2.62) | 3.78 (2.86)
    PCL - Cluster E Arousal | 12.88 (7.25) | 8.31 (6.34) | 10.59 (7.15)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms
Description: Self-report, measured by the PTSD checklist, civilian version (PCL-5). 20-item self-report questionnaire, assessed severity of symptoms that parallel the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) diagnostic criteria for PTSD. Participants were asked to indicate the extent to which they were bothered by problems experienced in the past month in relation to a traumatic experience of abuse or act of violence (0 = not at all to 4 = extremely). Total severity score (range: 0-80; higher scores indicating higher symptom severity, >= 33 indicating PTSD) and subscale totals (Avoidance - Cluster C, range: 0-8, higher scores indicating higher avoidance symptom severity; and Hyperarousal - Cluster E, range: 0-24, higher scores indicating higher hyperarousal symptom severity) were examined.
Time Frame: 90 Days, 180 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Health Treatment | Standard of Care
Number analyzed (Participants) | 32 | 32
score on a scale
  PCL - total symptom severity (3 mos) | 25.79 (5.40) | 23.04 (3.60)
  PCL - total symptom severity (6 mos) | 28.61 (5.04) | 22.50 (3.47)
  PCL - Cluster C Avoidance (3 mos) | 2.21 (0.63) | 2.23 (0.39)
  PCL - Cluster C Avoidance (6 mos) | 2.96 (0.60) | 2.71 (0.47)
  PCL - Cluster E Hyperarousal (3 mos) | 7.47 (1.36) | 8.00 (1.21)
  PCL - Cluster E Hyperarousal (6 mos) | 7.91 (1.54) | 6.75 (1.10)
Statistical Analysis 1: Comparison: Mental Health Treatment vs Standard of Care; Statistical analyses reported below is for PCL - Total at 3 months; Test type: Superiority — A sample size of 60 was chosen as adequate to examine the feasibility and acceptability of a pilot randomized controlled trial (RCT) with two conditions; p = 0.08, Mixed Models Analysis — A priori threshold for statistical significance was p<.05. The p-value presented corresponds to the time by condition interaction parameter; To assess changes in PTSD symptoms over time by intervention condition, linear mixed models were fit using the PROC MIXED procedure in SAS

2. Primary Outcome: HIV Medication Adherence (% Adherent)
Description: Assessed through biomarkers of dried blood spots (DBS) testing for presence of antiretroviral therapy (ART) (tenofovir, emtricitabine, and efavirenz) at 6 month assessment, supplemented by viral load (VL; considered adherent if VL <=40 copies/ml) when DBS unavailable. Outcome dichotomized.
Time Frame: 180 days
Population: Subset of participants newly initiating ART (excluding re-initiators and non-initiators; n=54, 49 with biomarker data)
Measure: Count of Participants; unit: Participants
Arm/Group | Mental Health Treatment | Standard of Care
Number analyzed (Participants) | 23 | 26
Participants | 19 | 15
Statistical Analysis 1: Comparison: Mental Health Treatment vs Standard of Care; Test type: Superiority — A sample size of 60 was chosen as adequate to examine the feasibility and acceptability of a pilot RCT with two conditions; p = 0.05, Chi-squared — A priori threshold was defined as p<0.05

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Mental Health Treatment | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02223390/Prot_SAP_000.pdf